CLINICAL TRIAL: NCT04057859
Title: A Prospective, Single Arm Study in Prostate Cancer Patients Managed With Androgen Deprivation Therapy to Examine the Effect of Nutritional Guidance and Aerobic/Resistance Fitness Training (ELIFIT)
Brief Title: PCa Patients Managed With ADT to Examine the Effect of Nutritional Guidance and Aerobic/Resistance Fitness Training
Acronym: ELIFIT
Status: Completed | Type: Observational
Sponsor: CMX Research (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: CMX-SC-2013-001
Record Dates: First submitted 2015-07-30; First posted 2019-08-15 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Cancer of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to examine the level of activity in the prostate cancer population treated with Androgen Deprivation Therapy (ADT).

DETAILED DESCRIPTION:
The aim of the current observational study will be to examine the level of activity in the prostate cancer population treated with ADT therapy; specifically, the impact of physical activity levels along with nutritional guidance through physician support. The application of an innovative technology to motivate patients will also be examined through the provision of an accelerometer/pedometer (NIKE+ FuelBand). The physical activity will be monitored by a NIKE+ Fuelband or tracked on an activity log.This study will assess the clinical and patient reported outcomes relevant to the management of their prostate cancer, in conjunction with a program assessing daily physical activities and nutritional guidance on the impact on the patient's quality of life, mobility and weight maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Male patient aged ≥ 18 years old
* Able to read and sign an approved Informed Consent Form (ICF)
* Diagnosed with locally advanced or metastatic prostate cancer
* Patient is treatment naive for ADT or has started ADT (3 or 4 month depot injection) AND has not received more than 1 treatment of 3 or 4 month ADT OR Patient is on intermittent therapy with an ADT agent and will be restarting ADT (3 or 4 month depot injection)
* ECOG (Eastern Cooperative Oncology Group) score of ≤ 2
* Willingness to track weekly physical activities with or without participating in a home based exercise program during the course of this study. The physical activities will be tracked with a weekly activity log or a NIKE+ Fuelband

Exclusion Criteria:

* Currently participating in a clinical study or observational study
* Has a survival expectancy of < 2 years
* Has any other condition that, in the opinion of the treating physician, may affect the patient's health or outcome of the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are being treated for prostate cancer with urologists in a community or academic/hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Changes in the patient quality of life (QoL) using the EORTC QLQ-C30 | Month 0 to Month 36
  The EORTC QLQ-C30 is a questionnaire designed to measure quality of life of cancer patient.
Changes in the patient quality of life (QoL) using the FACT-P | Month 0 to Month 36
  The FACT-P (Functional Assessment of Cancer Therapy - Prostate) is a questionnaire used to assess the health-related quality of life in men with prostate cancer.
Changes in the patient quality of life (QoL) using the FACIT Fatigue Scale | Month 0 to Month 36
  The FACIT (Functional Assessment of Chronic Illness Therapy) Fatigue Scale is a questionnaire that measures an individuals level of fatigue during their usual daily activities over the past week.

SECONDARY OUTCOMES:
Determine compliance of home-based exercises and regular physical activities | 3 Years
  To determine the compliance of home-based exercises and regular physical activities using a weekly activity log.
Determine the impact of exercise and physician support on activity levels | 3 Years
  To determine the impact of exercise and physician support on activity levels using the weekly activity log, home diary or NIKE+ Fuelband.
Assess the impact of nutritional guidance and exercise with physician support on BMI | 3 Years
  To determine if BMI (body mass index) scores decrease with nutritional guidance and exercise with physician support.
Mobility of prostate cancer patients measured by TUG Test | 3 Years
  To assess the impact of nutritional guidance and exercise with physician support on the mobility of prostate cancer patients treated with ADT as measured by the Timed Up and Go Test (TUG)
Determine the safety and tolerability of ADT in the management of prostate cancer | 3 Years
  Safety and tolerability will be assessed based on the number and type of adverse events collected over the study duration.
# of patients who discontinued prescribed treatment or intermittent usage of prescribed treatment | 3 Years
  To determine # of patients who discontinued ADT therapy over the course of the study with reasons describing why.
Mobility of prostate cancer patients measured by Five Times Sit to Stand Test (FTSST) | 3 years
  To assess the impact of nutritional guidance and exercise with physician support on the mobility of prostate cancer patients treated with ADT as measured by the Five Times Sit to Stand Test (FTSST).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Casey, MD, Study Director — CMX Research
Locations (23):
- Canada (23):
  - Southern Interior Medical Research Inc., Kelowna, British Columbia
  - Silverado Research Inc., Victoria, British Columbia
  - Barrie Urology Group, Barrie, Ontario
  - Euroscope Inc., Barrie, Ontario
  - Dr. Gregory Leal, Belleville, Ontario
  - Jonathan Giddens Medical Professional Corp., Brampton, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - Kenneth Jansz Medical Professional Corp., Burlington, Ontario
  - Michael L. Pianezza Medicine Professional Corp., Greater Sudbury, Ontario
  - Northern Urology Centre, Greater Sudbury, Ontario
  - Stanley Flax Medical Professional Corp., North York, Ontario
  - The Fe/Male Health Centres, Oakville, Ontario
  - The Fe/Male Health Centre, Oakville, Ontario
  - Kawartha Urology, Peterborough, Ontario
  - Urology Clinic, Scarborough Village, Ontario
  - Dr. Jonathan Chan Medical Professional Corp., Toronto, Ontario
  - Umesh Jain Medicine Professional Corp., Toronto, Ontario
  - Recherches Cliniques Theradev, Granby, Quebec
  - UroLaval, Laval, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Ultra-Med Inc., Pointe-Claire, Quebec
  - CHU de Quebec - L'hotel-dieu de Quebec, Québec, Quebec
  - Centre de Recherche en Urologie de Lanaudiere, Saint-Charles-Borromée, Quebec

IPD SHARING:
Plan to Share IPD: Undecided